CLINICAL TRIAL: NCT02786979
Title: Combination of Beraprost Sodium Tablets (Dorner) and Aspirin for Prevention of Arteriosclerosis Progress in Type 2 Diabetes Mellitus Patients
Brief Title: Efficacy and Safety of Dorner Tablets and Aspirin for Prevention of Arteriosclerosis Progress in Type 2 Diabetes Mellitus Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Upon interim analysis, sponsor's decision due to absence of demonstration of efficacy.
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DorDM002
Record Dates: First submitted 2016-05-26; First posted 2016-06-01 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Arteriosclerosis; beraprost; Aspirin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Arteriosclerosis | interventions — beraprost; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Beraprost sodium tablet and Aspirin combination group (Experimental): Oral
  Interventions: Drug: Beraprost; Drug: Aspirin
- Aspirin Group (Experimental): Oral
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Beraprost — Oral
  Other Names: Dorner (R)
  Arms: Beraprost sodium tablet and Aspirin combination group
Drug: Aspirin — Oral

SUMMARY:
The objective was to evaluate the efficacy and safety of combination of beraprost and aspirin for prevention of arteriosclerosis progress in type 2 diabetes mellitus patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as type 2 diabetes mellitus;
* Patients who had the intima-media thickness (IMT) of carotid artery ≥1.1 mm in at least one side;
* Patients who had results of aspartate aminotransferase, alanine aminotransferase, and serum creatinine no more than 1.5 times higher than the upper limit of normal;
* Patients who had not cardio or cerebral vascular events within 3 months, including non-fatal myocardial infarction, stable and unstable angina pectoris, and non-fatal cerebral ischemic and hemorrhagic stroke;
* Patients who had their systolic blood pressure <160 mmHg, diastolic blood pressure <100 mmHg, and glycated hemoglobin (HbA1c) <8.0%;
* Patients who had not taken any medications with antithrombotic and antiplatelet effect within 3 months;

Exclusion Criteria:

* Patients who had peptic ulcer or active alimentary tract hemorrhage;
* Patients who had a known allergy to prostacycline or non-steroid medications;
* Patients who were pregnant, breast feeding, or had planned to be pregnant;
* Patients who were attending or had attended any clinical studies within 3 months;

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2010-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in carotid intima-media thickness | Baseline to Year 3
Incidence and severity of treatment-emergent adverse events | Up to 3 years
Safety assessed by vital signs: body temperature | Up to 3 years
Safety assessed by vital signs: pulse rate | Up to 3 years
Safety assessed by vital signs: respiratory rate | Up to 3 years
Safety assessed by vital signs: blood pressure (systolic blood pressure and diastolic blood pressure) | Up to 3 years
Number of participants with abnormal laboratory values and/or adverse events related to treatment | Up to 3 years

SECONDARY OUTCOMES:
Death rate | Up to 3 years
Incidence of any vascular event | Baseline to Year 3
  Vascular events include sudden death, death caused by the vascular event, non-fatal coronary hear disease (CHD), non-fatal cerebrovascular diseases, and non-fatal aorta and peripheral artery disease (PAD)
Change from baseline in Ankle-brachial index | Baseline to Year 3
Change from baseline in Pulse wave velocity | Baseline to Year 3
Change from baseline in Oxidative stress indices | Baseline to Year 3
  Oxidative stress indices: superoxide dismutase and nitrotyrosine
Change from baseline in value of VCAM-1 | Baseline to Year 3
  VCMA-1: vascular cell adhesion molecule
Change from baseline in value of TNF-α | Baseline to Year 3
  TNF: tumor necrosis factor

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (6):
- China (6):
  - Site CN00001, Beijing, Beijing Municipality
  - Site CN00002, Beijing, Beijing Municipality
  - Site CN00004, Guangzhou, Guangdong
  - Site CN00003, Shanghai, Shanghai Municipality
  - Site CN00005, Chengdu, Sichuan
  - Site CN00006, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Undecided